CLINICAL TRIAL: NCT00968643
Title: A Randomised Phase III Trial of Two Fractionation Schemes in the Treatment of Malignant Spinal Cord Compression
Brief Title: Spinal Cord Compression. ICORG 05-03, V6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-03 ICORG; ICORG-05-03; EU-20952
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-08

CONDITIONS: Spinal Cord Compression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: spinal cord compression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Spinal Cord Compression | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (control) (Active Comparator): Patients undergo radiotherapy to the area of spinal cord compression once daily for 5 days (total of 20 Gy).
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo a single fraction of radiotherapy to the area of spinal cord compression (total of 10 Gy).
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Given in multiple fractions or as a single fraction

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known which radiation therapy schedule is more effective in treating patients with malignant spinal cord compression.

PURPOSE: This randomized phase III trial is studying two different radiation therapy schedules to compare their side effects and how well they work in treating patients with malignant spinal cord compression.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the response in patients with malignant spinal cord compression treated with single fraction (10 Gy) radiotherapy vs standard multiple fraction (20 Gy) radiotherapy.
* To compare the toxicity of these treatment regimens in these patients.

Secondary

* Examine the safety, practicability, and efficacy of treatment with a single 10 Gy fraction of radiotherapy in these patients.
* Analyze the initial neurological status, document the response to treatment, and calculate median survival of these patients.
* Perform an economic impact analysis comparing the two treatment arms.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients undergo radiotherapy to the area of spinal cord compression once daily for 5 days (total of 20 Gy).
* Arm II: Patients undergo a single fraction of radiotherapy to the area of spinal cord compression (total of 10 Gy).

Patients complete the EORTC QLQ-C30 quality-of-life questionnaire at baseline, at 5 weeks, and then every 3 months thereafter.

After completion of study treatment, patients are followed up at 1 and 5 weeks, at 3 months, and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, excluding the following:

  * Leukemia
  * Myeloma
  * Germ cell tumor
  * Primary tumor of the spine or vertebral column
* Diagnosis of malignant spinal cord compression confirmed by MRI of the entire spine
* Deemed inoperable or unsuitable for neurosurgical intervention at the time of initial assessment
* No single bone metastasis with controlled primary site

PATIENT CHARACTERISTICS:

* Karnofsky performance status 30-100%
* No medical or psychiatric condition that, in the opinion of the investigator or research team, would contraindicate study participation

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the involved area of the spinal cord such that further treatment exceeds spinal cord tolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2006-01; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mobility status: measured by the change in mobility status between baseline and 5 weeks, as measured by the in-house mobility scale | 5 weeks from date of randomisation

SECONDARY OUTCOMES:
Quality of life as assessed by the EORTC QLQ-C30 version 3 quality-of-life questionnaire | 5 weeks from date of randomisation
Toxicity: assessed at first follow-up, evaluated as per standard RTOG acute and long-term toxicity scale | 1 week after completion of therapy
Pain control: assessed using a Visual Analogue Scale | Until death
Overall survival: the survival duration will be calculated from time of randomisation to death whatever cause | Until death
Sphincter function: assessed using an 'In-House' Bladder Function Scale | Until death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, Principal Investigator — St Luke's Radiation Oncology Network
Locations (4):
- Ireland (4):
  - Cork University Hospital, Cork
  - Saint Luke's Radiation Oncology Network (SLRON), Dublin
  - Galway University Hospital, Galway
  - Whitfield Cancer Centre at Whitfield Clinic, Waterford

REFERENCES:
- [Derived] Thirion PG, Dunne MT, Kelly PJ, Flavin A, O'Sullivan JM, Hacking D, Sasiadek W, Small C, Pomeroy MM, Martin J, McArdle O, Parker I, O'Sullivan LS, Shannon AM, Clayton-Lea A, Collins CD, Stevenson MR, Alvarez-Iglesias A, Armstrong JG, Moriarty M. Non-inferiority randomised phase 3 trial comparing two radiation schedules (single vs. five fractions) in malignant spinal cord compression. Br J Cancer. 2020 Apr;122(9):1315-1323. doi: 10.1038/s41416-020-0768-z. Epub 2020 Mar 11. PMID 32157242